CLINICAL TRIAL: NCT00293852
Title: Collaborative Care for Heart Failure Patients With the Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Allison Pritchett, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-18155
Record Dates: First submitted 2006-02-17; First posted 2006-02-20 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Heart Failure, Congestive; Metabolic Syndrome X
Keywords: Heart failure, Congestive; Metabolic Syndrome X; Ambulatory Care; Health behavior
MeSH Terms: conditions — Heart Failure; Metabolic Syndrome; Health Behavior

ARMS (2):
- Usual Care (No Intervention)
- Collaborative Care (Experimental)
  Interventions: Procedure: Outpatient clinic follow-up

INTERVENTIONS:
Procedure: Outpatient clinic follow-up
  Arms: Collaborative Care

SUMMARY:
Heart failure is a condition where the heart does not pump enough blood to the rest of the body. People with heart failure may have another condition called the "metabolic syndrome"( having excess fat in the belly, high blood pressure, high fat in the blood, low level of good cholesterol and high blood sugar). People who have both heart failure and the metabolic syndrome often see many doctors. A new clinic has been formed at Ben Taub General Hospital that includes a specialist in heart failure (cardiologist) and in the metabolic syndrome (endocrinologist) as well as patient teaching. The goal of this study is to randomize patients with the metabolic syndrome who are admitted to the hospital for heart failure to this clinic (collaborative care) versus the usual doctor appointments (usual care). The purpose of this study is to see if collaborative care is better medical care than usual care. Specifically, we will see if patients in collaborative care will have:

1. fewer admissions to hospitals for illness
2. better blood pressure, sugar, fat and heart failure control
3. better patient satisfaction and knowledge about their diseases
4. lower levels of inflammation.

DETAILED DESCRIPTION:
A striking feature of the Harris County Hospital District heart failure population is that the prevalence of obesity (50.8%) and the metabolic syndrome (48.9%) exceeds that of the general U.S. population. The metabolic syndrome is defined as the presence of 3 out of 5 components: abdominal obesity, elevated blood pressure, dyslipidemias (↑ triglycerides and ↓ high density lipoprotein) and insulin resistance and hyperglycemia. Current treatment recommendations for the metabolic syndrome include lifestyle modification (diet, exercise, and weight control) and targeted pharmaceutical therapy for the individual components. Although specialized care for the metabolic syndrome has not been reported, separately, both specialty heart failure care and endocrinology care have been shown to reduce hospital admissions and health care costs, increase target medication titration and disease control, improve quality of life, and survival in patients with heart failure and diabetes respectively. As both heart failure and the metabolic syndrome are commonly found in the same patients, collaborative out-patient management of both conditions in the same clinic is novel and may have a significant impact on outcomes.

Hypothesis:

Compared to usual post-discharge follow-up, collaborative treatment of heart failure patients with the metabolic syndrome by a team composed of an endocrinologist, cardiologist, patient educator, nurse and case manager will result in:

* Decreased hospital readmissions and emergency room visits
* Health care cost savings
* Increased achievement of treatment goals (target blood pressure, HgbA1c, lipids, and heart failure medication titration)
* Improved patient satisfaction, knowledge, and compliance
* Lower levels of markers of inflammation and insulin resistance

ELIGIBILITY:
Inclusion Criteria:

* Individuals with heart failure of ischemic or non-ischemic etiologies
* Age ≥18 years
* Admitted to the hospital with a primary diagnosis of heart failure (need not be their first admission for heart failure)
* Meets the modified Framingham criteria for the diagnosis of heart failure (2 major OR 1 major / 2 minor are required):

MAJOR: paroxysmal nocturnal dyspnea (sudden shortness of breath at night), orthopnea (shortness of breath when supine), elevated jugular venous pressure, rales, the presence of an S3 heart sound, cardiomegaly on chest X-ray, pulmonary edema on chest X-ray

MINOR: lower extremity edema, night cough, dyspnea on exertion, hepatomegaly, pleural effusion on chest X-ray, heart rate > 120 bpm, weight loss > 10 pounds in 5 days while in hospital

• Meets the National Cholesterol Education Panel criteria for the metabolic syndrome (3 of 5 criteria must be present):

* waist > 40 in for men, 35 in for women
* blood pressure ≥ 130/85 mmHg or hypertension
* triglycerides ≥150 mg/dL
* fasting glucose ≥ 100 mg/dL or diabetes
* high density lipoprotein level (HDL) < 40 mg/dL for men, <50 for women

Exclusion Criteria:

Patients will be excluded if they do not meet the definitions for heart failure and the metabolic syndrome listed above. Also, heart failure patients admitted for a diagnosis other than acute heart failure exacerbation will not be included. Other exclusion criteria include:

* A condition, other than heart failure, that limits a patient's survival (such as cancer, active hepatitis, advanced HIV infection etc.)
* Factors that may limit adherence to interventions or affect conduct of the trial

  * Unable or unwilling to given informed consent
  * Mental incapacity that limits patient's ability to live independently and benefit from patient education

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2006-02; Primary Completion 2009-10-14 (Actual); Study Completion 2015-12-10 (Actual)

PRIMARY OUTCOMES:
the number of rehospitalizations and emergency room visits for heart failure exacerbation | 1 year

SECONDARY OUTCOMES:
health care costs | 1 year
the achievement of goal doses of heart failure medications and target measures of the metabolic profile | 1 year
the change in levels of insulin resistance and inflammatory biomarkers | 1 year
overall patient satisfaction, disease understanding, and "self-management" skills | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Allison M. Pritchett, M.D., Principal Investigator — Baylor College of Medicine; Ramaswami Nalini, M.B.B.S, Principal Investigator — Baylor College of Medicine; Ashok Balasubramanyam, M.D., Principal Investigator — Baylor College of Medicine
Locations (1):
- Ben Taub General Hospital, Houston, Texas, United States